CLINICAL TRIAL: NCT00407069
Title: Role of Antimicrobial Peptides in Host Defense Against Vaccinia Virus (ADVN AMP01)
Brief Title: Role of Antimicrobial Peptides in Host Defense Against Vaccinia Virus
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ADVN AMP 01
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and skin samples will be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Active Atopic Dermatitis (AD): Pediatric and adult subjects who fulfill the criteria for AD, a chronic inflammatory skin disease.
- Inactive Atopic Dermatitis (AD): Adult subjects with a prior history of active AD that has been quiescent for at least 1 year.
- Psoriatics: Adult subjects who fulfill the criteria for plaque psoriasis, a chronic inflammatory skin disease.
- Asthmatics (without a history of AD): Adult subjects who fulfill the criteria for asthma (reactive airway disease) and have a negative history of skin disease.
- Eczema Herpeticum (EH: Pediatric and adult AD subjects with a history of EH.
- Healthy Volunteers: Healthy individuals with no history of skin or respiratory disease.

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disorder characterized by recurrent viral skin infections. Recent studies have demonstrated that the skin of people with AD my have decreased antimicrobial peptide (AMP) expression. The purpose of this study is to compare smallpox virus replication and the number of AMPs and other antiviral molecules in people with AD, as compared to those seen in people with psoriasis or asthma, or healthy individuals.

DETAILED DESCRIPTION:
AD is a chronic inflammatory skin disease characterized by frequent viral skin infections. Recent studies have found that components in the skin of people with AD may block AMP expression. AMPs are responsible for preventing infection from viruses. The purpose of this study is to examine smallpox virus replication and AMP expression in the skin of patients with AD as well as identify other antiviral molecules involved in immune response. These findings will be compared with those of people with psoriasis or asthma, or healthy individuals. This study will consist of one study visit at which skin and blood samples will be taken.

ELIGIBILITY:
Inclusion Criteria for Participants With AD:

* 2 years of age or older
* History of active or inactive AD OR eczema herpeticum, as defined by the ADVN standardized diagnostic criteria
* Parent or guardian willing to provide informed consent, if applicable
* Male or female of any race and ethnicity

Inclusion Criteria for Participants With Asthma or Psoriasis, and for non-atopic controls:

* 18 years or older
* History of psoriasis OR history of asthma not requiring systemic medications
* Parent or guardian willing to provide informed consent, if applicable
* Male or female of any race and ethnicity

Exclusion Criteria:

* Oral corticosteroids or any systemic immunosuppressive or immunomodulatory medication within 28 days prior to study entry
* Immunotherapy within 3 months prior to study entry
* History of bleeding disorder
* Aspirin, oral antihistamines, oral antibiotics, oral cyclosporine, or topical medications within 7 days of screening visit including, but not restricted to, Protopic, Elidel, topical corticosteroids, and topical antibiotics
* Anxiolytic agents and antidepressants within 2 days of screening visit
* Diabetic requiring medication
* Autoimmune or immunodeficiency
* Active fungal, bacterial, or viral infections within 7 days prior to study entry
* Active systemic cancer. Participants with uncomplicated nonmelanoma skin cancer are not excluded.
* Theophylline or leukotriene antagonists within 24 hours of screening visit
* Received any vaccination within 30 days prior to study entry
* Known lidocaine allergy
* Previously vaccinated for smallpox
* Pregnant or breastfeeding

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People of good general health
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2005-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Expression of vaccinia virus mRNA in non-lesional skin following inoculation with untreated vaccinia virus will be evaluated using real-time RT-PCR (Reverse transcription polymerase chain reaction). | 5 years

SECONDARY OUTCOMES:
Expression of cytokines, AMPs, other antiviral molecules, or epidermal differentiation proteins in non-lesional skin prior to and after inoculation with vaccinia virus will be evaluated using real-time RT-PCR. | 5 years
Keratinocytes will be stimulated with vaccinia virus in the presence and absence of Th1 or Th2 cytokines. Non-lesional AD skin will be stimulated with vaccinia virus in the presence of antibodies that neutralize Th2 cytokines. | 5 years
Vaccinia virus replication will be evaluated using a standard viral plaque assay in BS-C-1 cells and by analyzing vaccinia virus mRNA expression using real-time RT-PCR in keratinocytes and BS-C-1 cells. | 5 years
Expression of over 20,000 genes will be evaluated by GeneChip microarrays in non-lesional skin, and PBMCs stimulated with vaccinia virus. Real-time RT-PCR of skin and PBMC will be used to confirm gene alterations found in GeneChip microarrays. | 5 years
Ability of structural analogues of CSAs (Cyclosporine) to kill purified vaccinia virus as well as keratinocytes infected with vaccinia virus in vitro. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Howell MD, Jones JF, Kisich KO, Streib JE, Gallo RL, Leung DY. Selective killing of vaccinia virus by LL-37: implications for eczema vaccinatum. J Immunol. 2004 Feb 1;172(3):1763-7. doi: 10.4049/jimmunol.172.3.1763. PMID 14734759
- [Background] Nomura I, Goleva E, Howell MD, Hamid QA, Ong PY, Hall CF, Darst MA, Gao B, Boguniewicz M, Travers JB, Leung DY. Cytokine milieu of atopic dermatitis, as compared to psoriasis, skin prevents induction of innate immune response genes. J Immunol. 2003 Sep 15;171(6):3262-9. doi: 10.4049/jimmunol.171.6.3262. PMID 12960356
- [Background] Howell MD, Wollenberg A, Gallo RL, Flaig M, Streib JE, Wong C, Pavicic T, Boguniewicz M, Leung DY. Cathelicidin deficiency predisposes to eczema herpeticum. J Allergy Clin Immunol. 2006 Apr;117(4):836-41. doi: 10.1016/j.jaci.2005.12.1345. Epub 2006 Feb 14. PMID 16630942
- [Background] Leung DY, Boguniewicz M, Howell MD, Nomura I, Hamid QA. New insights into atopic dermatitis. J Clin Invest. 2004 Mar;113(5):651-7. doi: 10.1172/JCI21060. PMID 14991059
- [Result] Howell MD, Gallo RL, Boguniewicz M, Jones JF, Wong C, Streib JE, Leung DY. Cytokine milieu of atopic dermatitis skin subverts the innate immune response to vaccinia virus. Immunity. 2006 Mar;24(3):341-8. doi: 10.1016/j.immuni.2006.02.006. PMID 16546102
- [Result] Howell MD, Gao P, Kim BE, Lesley LJ, Streib JE, Taylor PA, Zaccaro DJ, Boguniewicz M, Beck LA, Hanifin JM, Schneider LC, Hata TR, Gallo RL, Kaplan MH, Barnes KC, Leung DY. The signal transducer and activator of transcription 6 gene (STAT6) increases the propensity of patients with atopic dermatitis toward disseminated viral skin infections. J Allergy Clin Immunol. 2011 Nov;128(5):1006-14. doi: 10.1016/j.jaci.2011.06.003. Epub 2011 Jul 18. PMID 21762972
- [Result] Grigoryev DN, Howell MD, Watkins TN, Chen YC, Cheadle C, Boguniewicz M, Barnes KC, Leung DY. Vaccinia virus-specific molecular signature in atopic dermatitis skin. J Allergy Clin Immunol. 2010 Jan;125(1):153-159.e28. doi: 10.1016/j.jaci.2009.10.024. PMID 20109744
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY10 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY10 — ImmPort study identifier is SDY10.
- Available data/document: Study Protocol: SDY10 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY10 — ImmPort study identifier is SDY10.
- Available data/document: Study design, -summary, -files; participant demographics, et al.: SDY10 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY10 — ImmPort study identifier is SDY10.